CLINICAL TRIAL: NCT03548428
Title: Randomized Phase II, 2-arm Study of Immunomodulation with Atezolizumab Concomitant with High Dose Radiation (SBRT) Versus SBRT Alone in Patients with Oligometastatic Sarcomas
Brief Title: Stereotaxic Body Irradiation of Oligometastase in Sarcoma (Stereosarc)
Acronym: Stereosarc
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Collaborators: Centre Hospitalier Universitaire de Caen (Other); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017_16
Record Dates: First submitted 2018-01-31; First posted 2018-06-07 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Sarcoma; Radiosurgery
Keywords: Atezolizumab; Oligometastatic Sarcomas; stereotactic body radiation therapy
MeSH Terms: conditions — Sarcoma | interventions — atezolizumab; Radiation

STUDY DESIGN:
Intervention Model Description: Open label, Phase II, prospective, multicentric, randomized study 2:1, 2 arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Experimental): SBRT + Atezolizumab
  Interventions: Drug: Atezolizumab; Radiation: SBRT
- B (Active Comparator): SBRT
  Interventions: Radiation: SBRT

INTERVENTIONS:
Drug: Atezolizumab — 1200mg IV every 3 weeks for 4 months
  Arms: A
Radiation: SBRT — 3 to 5 fractions depending on tumor size
  Other Names: High Dose Radiation

SUMMARY:
Up to 50% of soft tissue sarcoma (STS) patients will develop metastases in the course of their disease. Cytotoxic therapy is a standard treatment in this setting but yields average tumor response rates of 25% at first line and ≤10% at later lines. It is also limited in the number of lines and courses by tolerance issues. Trials include poly/oligometastases indistinctively and suggest that consolidation ablation is used in ~20% of patients with residual oligometastases refractory to chemotherapy. Oligometastases represent a stage of disease between completely absent and widely metastatic, and which might be cured if the limited numbers of metastatic sites are eradicated. Ablative strategies to treat patients with oligometastases from sarcomas yield prolonged survival times and stereotactic body radiation therapy (SBRT) is associated with excellent tolerance. Surgery may be offered in selected metastatic cases. Alternatively and increasingly, SBRT yields high control rates at treated sites (≥ 80%). The so-called radioresistance of sarcomas is overcome by the high doses per fraction made possible owing to the high precision achieved with SBRT. SBRT is an accepted treatment strategy provided that tumor burden remains limited in the number and size of metastases. Systemic treatment can be combined with SBRT. SBRT may produce abscopal effects where tumors outside the irradiation area also demonstrate tumor shrinkage in some occurrences. SBRT produces systemic antitumoral immune response in certain conditions and enhances radiation-induced tumor cell death compared to conventional lower dose irradiation. Abscopal effects have been potentialized with SBRT/immunotherapy in several tumor models. Sarcomas are a privileged target tumor given their high metastatic propensity.

Several potent immunomodulators that skew the tumor immune microenvironment toward a proimmunity context are being investigated in STS either alone or in combination with chemotherapy or targeted therapy. The PD-1 receptor is present within the tumor microenvironment, and limits the activity of infiltrating cytotoxic T lymphocytes, thus blocking effective immune responses. The action of PD-1 is triggered upon binding to its ligands. PD-1 can stimulate the immunosuppressive function of regulatory T cells. Moreover, blockade of PD-1 can stimulate anti-tumor immune responses. Significant responses have been obtained in several sarcomas with acceptable tolerance. Preliminary clinical experience suggests that immunotherapy can be efficient in refractory leiomyosarcomas. Several drugs targeting the PD-1/PD-L1/2 axis are ongoing either as single agents or in combination with ipilimumab, kinase inhibitors, or chemotherapy in STS subtypes. Combination of radiotherapy with immunotherapy is included as a means of increasing tumor antigen release in metastatic STS. Immunomodulated SBRT is a particularly attractive strategy, given the potential of radiation to induce cytotoxicity in tumors and induce abscopal effects. A phase II radiation trial showed increased apoptosis-, intra-tumoral dendritic cells and accumulation of intratumoral T cells in STS with correlation with tumor-specific immune responses.

We here propose a randomized phase II study to prolong progression-free survival (PFS) with the combination of SBRT/immunotherapy in oligometastatic STS patients.

SBRT is well-tolerated with hardly any severe toxicity (fewer than 5% acute and late grade 3 toxicities). It is performed in an ambulatory setting in only a few treatment fractions. Associations between irradiation and immunomodulatory agents appear to be synergistic and show favorable tolerance profiles. Immunomodulatory agents have a more favorable toxicity profile than cytotoxic agents with about 65% overall acute toxicities. Immunotherapy selectively binds to PD-L1 and competitively blocks its interaction with PD-1.

Compared with anti-PD-1 antibodies that target T-cells, immunotherapy targets tumor cells, and is therefore may induce fewer side effects, including a lower risk of autoimmune-related safety issues, as blockade of PD-L1 leaves the PD-L2 - PD-1 pathway intact to promote peripheral self-tolerance.

Stereotactic irradiation is associated with an excellent tolerance with rates of grade 3 or more toxicities below 5%.

Preliminary data of toxicity with the association of stereotactic irradiation and immunotherapy show no cumulative toxicity in association with immunotherapy. However, their incidence and characteristics are no different from that observed with stereotactic irradiation alone. Moreover, intracranial metastases are exceptional in sarcomas.

The toxicity of the association for extracranial stereotactic irradiation does not seem to be increased either.

DETAILED DESCRIPTION:
Open label, Phase II, prospective, multicentric, randomized study 2:1, 2 arm study designed to evaluate the efficacy of a Stereotactic Body Radiation Therapy treatment associated with immunotherapy versus a Stereotactic Body Radiation Therapy treatment only.

Primary objective The primary objective is to evaluate the efficacy, in term of progression-free survival (PFS) rate at 6 months, of immunomodulated stereotactic irradiation in oligometastatic sarcoma patients.

Secondary Objectives

* PFS by immune response criteria.
* ratio PFS after radiotherapy/PFS during the previous line of treatment
* Objective response rate.
* Rate of progression-free survival (PFS) at 6 months by line of treatment and histology.
* Evaluation of the toxicity of the treatment.
* Overall survival.
* Evaluation of the quality of life of patient treated by the combination of radio- and immunotherapy or radiotherapy only.
* Evaluation of the cost of treatment.
* Rate of PET-CT at inclusion
* Correlative study: Impact of biomarkers on clinical endpoints.
* Developing a mathematical models for STS treatment by SBRT + immunotherapy predictive of oligo versus poly metastatic evolution

The treatment to be used in this study is the Atezolizumab concomitant with High Dose Radiation (SBRT) or the SBRT Alone Atezolizumab Subjects randomized in the experimental arm will receive Atezolizumab 1200 mg in combination with SBRT, Q3W (6 cycles) for 4 months until progression/completion. The Atezolizumab will be provided by the Sponsor (Centre Antoine Lacassagne).

Chemotherapy will be discontinued in case of progression, unacceptable toxicity, or withdrawal of patient consent to receive study treatment.

Radiation therapy SBRT can be performed with different equipments (CyberKnife, Truebeam, etc.). Adequate tumor tracking and patient setup/repositioning as well as online IGRT (image-guided radiation therapy) must be performed at each fraction. The maximal cumulative tumor diameter is 6 cm to maintain an advantageous risk-benefit ratio with SBRT. Two types of fractionation are proposed to account for tumor size and proximity of the tumor to sensitive organs at risk. Three fractions are proposed in favorable cases, 5 in more delicate cases. Fractions can be performed on consecutive days. Depending on cases, they may be delivered every other day; the whole SBRT duration should not exceed 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* • STS (leiomyosarcomas uterine/extra-uterine, liposarcomas, undifferentiated sarcomas), any grade

  * Progressive disease according to RECIST 1.1 criteria,
  * Metastatic disease (1-5 synchronous macroscopic metastases by chest and abdominopelvic CT, maximal cumulated diameter 10 cm); any anatomic site
  * First or second metastatic line
  * Be ≥ 18 years of age on day of signing informed consent.
  * Have a performance status of 0 or 1 on the ECOG Performance Scale.
  * Have at least one lesion mesurable by RECIST 1.1 for irradiation with a size of < 5 cm.
  * Demonstrate adequate organ function: Absolute neutrophil count (ANC) ≥1,500 /mcL; Platelets ≥100,000 / mcL; Hemoglobin ≥9 g/dL or ≥5.6 mmol/L; Serum creatinine ≤1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥50 mL/min for subject with creatinine levels > 1.5 X institutional ULN; Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN; AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases. All screening labs should be performed within 15 days of treatment initiation.
  * Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
  * Surgical ablation (or other ablative methods such as thermal ablative methods) remains possible if needed before SBRT, at least 4 weeks before randomisation and provided that at least one lesion needs to be treated by SBRT.
  * FFPE Tumor tissue collected before SBRT is available for immunohistochemistry (optional)
  * Archival metastatic biopsy blocks (or slides) on paraffin embedded samples available. If no archival material is available, a fresh biopsy should be performed if possible.
  * Be willing and able to provide written informed consent/assent for the trial.
  * affiliated with a health insurance system.

Exclusion Criteria:

* Is currently participating in, or has participated in, a study of an investigational agent or using an investigational device within 4 weeks prior to randomisation.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has had a prior monoclonal antibody within 4 weeks prior to randomisation or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy or targeted small molecule therapy within 4 weeks prior to randomisation or who has not recovered (i.e. ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent (Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study). If subjects received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Have had previous radical radiation to any tumour site within 4 weeks prior to randomisation
* Have had previous ablative treatment within 4 weeks prior to randomisation (radiofrequency, surgery)
* Has a tumour within 5 mm of the spinal cord (owing to rare reported cases of flare-up after initiation of immunotherapy)
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjögren's syndrome will not be excluded from the study.
* Has evidence of symptomatic interstitial lung disease or an active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance-abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g. HBsAg reactive) or Hepatitis C (e.g. HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* Has had major surgery or major blood transfusions (>3 packed cells) in the past 3 months.
* Receives IL-2, interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigational therapies; or chronic use of systemic corticosteroids (used in the management of cancer or non-cancer-related illnesses)
* Under-age patients
* Patients unable to express their consent
* Vulnerable persons as defined by article L1121-5 - 8:
* Pregnant women, women in labor or breast-feeding mothers, persons deprived of their freedom by judicial or administrative decision, persons hospitalized without their consent by virtue of articles L. 3212-1 and L. 3213-1 and who are not subject to the provisions of article L. 1121-8
* Persons admitted to a social or health facility for reasons other than research
* Adults subject to a legal protection order or unable to give their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2031-02-04 (Estimated)

PRIMARY OUTCOMES:
efficacy, in term of progression-free survival (PFS) rate at 6 months | 6 months
  Rate of progression-free survival (PFS)

SECONDARY OUTCOMES:
PFS by immune response criteria. | 5 years
  PFS by immune response criteria defined as the time between the date of randomizationrandomisation and the date of progression or the date of death or the date of last news.
ratio PFS after radiotherapy/PFS during the previous line of treatment | 5 years
  ratio PFS after radiotherapy/PFS during the previous line of treatment
Objective response rate. | 5 years
  Objective response rate defined according to RECIST criteria version 1.1
Rate of progression-free survival (PFS) at 6 months by line of treatment and histology. | 6 months
  Rate of progression-free survival (PFS) at 6 months as defined in the primary endpoint by line of treatment and by histology
Evaluation of the toxicity of the treatment | 6 months
  Toxicity will be graded according to National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4.0. The rate of grade ≥ 3 toxicities will be evaluated.
Overall survival | 5 years
  Overall Survival defined as the time between the date of randomizationrandomisation and the date of death or the date of last news for those still alive at the end of the follow-up.
Evaluation of the quality of life of patient treated by the combination of radio- and immunotherapy or radiotherapy only | 2 years
  Quality of life will be measured using standard quality of life questionnaire EORTC QLQc30
Evaluation of the cost of treatment | 4 months
  The cost of the treatment will be calculated on the basis of the length of hospitalization in days
Rate of PET-CT at inclusion | Baseline
  Rate of PET-CT scan performed at inclusion
Impact of biomarkers on PFS. | baseline, 6 months, at relapse within 5 years
  Impact of biomarkers (PD1/PDL1 immunostaining in tumor and microenvironment, CRP, albumin, neutrophils/lymphocytes at baseline and ctDNA at baseline, 6 months and relapse) on pfs
Impact of biomarker on response rate. | baseline, 6 months, at relapse within 5 years
  Impact of biomarkers (PD1/PDL1 immunostaining in tumor and microenvironment, CRP, albumin, neutrophils/lymphocytes at baseline and ctDNA at baseline, 6 months and relapse) on response rate
Developing a mathematical models for STS treatment by SBRT + immunotherapy predictive of oligo versus poly metastatic evolution | 5 years
  Validation of the predictive models

CONTACTS AND LOCATIONS:
Overall Officials: Juliette THARIAT, MD, Principal Investigator — Centre Hospitalier Universitaire de Caen
Locations (17):
- France (17):
  - Institut Bergonié, Bordeaux
  - Centre François BACLESSE, Caen
  - Centre Georges François LECLERC, Dijon
  - Centre Oscar LAMBRET, Lille
  - Centre Léon BERARD, Lyon
  - AP-HM CHU La Timone, Marseille
  - Institut Paoli CALMETTES, Marseille
  - Institut de cancérologie de Montpellier, Montpellier
  - Centre Antoine LACASSAGNE, Nice
  - APHP La Pitié, Paris
  - CHU de Poitiers, Poitiers
  - Centre Eugene MARQUIS, Rennes
  - Centre Henri BECQUEREL, Rouen
  - Institut de cancérologie Strasbourg Europe, Strasbourg
  - Institut Claudius REGAUD, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave ROUSSY, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] le Guevelou J, Debaigt C, Saada-Bouzid E, Viotti J, Khalladi N, Thibouw D, Penel N, Sunyach MP, Moureau-Zabotto L, Benchalal M, Veresezan O, Ducassou A, le Pechoux C, Jolnerovski M, Bazille C, Vaur D, Escande A, Serre R, Lovera C, Thariat J. Phase II study of concomitant radiotherapy with atezolizumab in oligometastatic soft tissue sarcomas: STEREOSARC trial protocol. BMJ Open. 2020 Sep 23;10(9):e038391. doi: 10.1136/bmjopen-2020-038391. PMID 32967883